CLINICAL TRIAL: NCT01681654
Title: Exercise and Nutrition for Head and Neck Cancer Patients: A Patient Oriented, Clinic-Supported Randomized Controlled Trial
Brief Title: Exercise and Nutrition for Head and Neck Cancer Patients
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Cancer Foundation (Other)
Responsible Party: Principal Investigator, Dr. Nicole Culos-Reed, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ENHANCE10001991
Record Dates: First submitted 2012-08-31; First posted 2012-09-10 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Cancer of Head and Neck
Keywords: Head/Neck Cancer; Exercise; Progressive Strength Training; Quality of Life; Cancer; Randomized Controlled Trial; Nutrition; Lifestyle Intervention
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Immediate Lifestyle Intervention - Maintenance Program (Experimental): Patients will receive a 12-week lifestyle program during treatment. Patients will also receive maintenance support following the 12-week program.
  Interventions: Behavioral: Lifestyle Intervention; Behavioral: Maintenance Intervention
- Immediate Lifestyle Intervention - No Maintenance Program (Experimental): Patients will begin the 12-week lifestyle intervention during treatment. Patients will not receive a maintenance support following the 12-week intervention.
  Interventions: Behavioral: Lifestyle Intervention
- Delayed Lifestyle Intervention - Maintenance Program (Experimental): Patients will receive a 12-week lifestyle intervention program following treatment (12 weeks after diagnosis). Patients will then receive maintenance support following the 12-week program.
  Interventions: Behavioral: Lifestyle Intervention; Behavioral: Maintenance Intervention
- Delayed Lifestyle Intervention - No Maintenance Program (Experimental): Patients will receive a 12-week lifestyle intervention program following treatment completion (12 weeks following diagnosis). Patients will not receive maintenance support following the 12-week program.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Participants in the Lifestyle Intervention will receive a 12-week individualized exercise and dietary program based on their exercise assessment and dual energy x-ray absorptiometry (DXA) scan results, will attend twice weekly group exercise classes, and perform their individualized at-home program an additional two times per week. In addition, participants will be required to attend six education sessions during the 12-week intervention.
Behavioral: Maintenance Intervention — Patients randomized to receive the Maintenance Program Intervention following treatment will receive a Survivorship Care Plan outlining their physical activity, dietary, and health behaviour progress throughout the program, future goals, individualized maintenance strategies, and optional drop-in exercise sessions.
  Arms: Delayed Lifestyle Intervention - Maintenance Program; Immediate Lifestyle Intervention - Maintenance Program

SUMMARY:
Research on physical activity and nutrition interventions aimed at positively impacting symptom management, treatment-related recovery and quality of life has largely excluded head and neck cancer populations. This translates into a lack of clinical programming available for these patient populations. Head and neck cancer patients deal with severe weight loss, with upwards of 70% attributed to lean muscle wasting, leading to extended recovery times, decreased quality of life (QoL), and impaired physical functioning. To date, interventions to address body composition issues have focused solely on diet, despite findings that nutritional therapy alone is insufficient to mitigate changes. A combined physical activity and nutrition intervention, that also incorporates important educational components known to positively impact behaviour change, is warranted for this population. Pilot work suggests that there is large patient demand and clinic support from the health care professionals for a comprehensive program. Therefore, the purpose of the present study is to examine the impact of timing of a 12-week PA and nutrition intervention (either during or following treatment) for HN cancer patients on body composition, recovery, serum inflammatory markers and quality of life. In addition, the investigators will examine the impact of a 12-week maintenance program, delivered immediately following the intervention, on adherence, patient-reported outcomes (i.e., management of both physical and psychosocial treatment-related symptoms and side-effects), as well as return to work. The investigators hypothesize that (1) patients who are randomized to the intervention at treatment start will experience improved symptom management and decreased lean body composition changes, directly improving recovery and QoL; (2) patients who receive a maintenance support program will have better long-term adherence and therefore superior treatment-related symptom management, physical and psychosocial functioning; and (3) return to work indices will improve and healthcare utilization costs will be lower in the participants who receive the immediate intervention (vs. delayed) as well as in those who receive the maintenance program (vs. no maintenance). This research will facilitate advancements in patient wellness, survivorship, and autonomy, and carve the path for a physical activity and wellness education model that can be implemented in other cancer centers.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 Years of Age
* Has received a diagnosis of nasopharyngeal, oropharyngeal or hypopharyngeal cancer
* Will receive radiation as part of treatment plan
* Able to walk without assistance
* Received clearance for exercise from treating oncologist
* Lives in Calgary, Alberta area
* Can speak and write English
* Is interested in participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Body Composition | At baseline (diagnosis), and then at 3, 6, 9 and 12 months post diagnosis
  DXA Scan will be used to assess body composition

SECONDARY OUTCOMES:
Quality of Life | At baseline (diagnosis), and then at 3, 6, 9 and 12 months post diagnosis
  Quality of Life will be assessed using the Functional Assessment of Cancer Therapy- Anemia module (FACT-AN), and the NCCN-FACT Fact Head/Neck Symptom Index-22 (FHNSI-22).
Physical Activity Behaviour | At baseline (diagnosis), and then at 3, 6, 9 and 12 months post diagnosis
  Physical activity will be assessed using Godin's (Godin, 1985) leisure score index (LSI) of the GLTEQ (Godin Leisure Time Exercise Questionnaire).
Smoking History | At baseline (diagnosis), and then at 3, 6, 9 and 12 months post diagnosis
  Smoking history will be assessed by a self report questionnaire which will classify patients as non-smokers, former smokers and current smokers.
Depression | At baseline (diagnosis), and then at 3, 6, 9 and 12 months post diagnosis
  Depression will be assessed using the Center for Epidemiological Studies on Depression Scale (CES-D).
Karnofsky Performance Score (KPS) | At baseline (diagnosis), and then at 3, 6, 9 and 12 months post diagnosis
  The Karnofsky Performance Score (KSP) will be used to measure the participant's general ability to accomplish tasks of daily-living and overall well-being.
Inflammatory Markers | At baseline (diagnosis), and then at 3, 6, 9 and 12 months post diagnosis
  Inflammatory factors will be evaluated as they are associated with cancer cachexia and muscle wasting and may be modified by exercise (Seruga et al., 2008; Baldwin, 2011). An overnight fasted blood draw will be collected at baseline, 3 months post diagnosis, 6 months post diagnosis, 9 months post diagnosis, and 12 months post diagnosis. Serum inflammatory cytokine concentrations will be assessed in-house (Dr. Raylene Reimer's laboratory) according to our established protocols. TNF, IL-6, IL-1, IL-8 and C-reactive protein will be quantified using Milliplex Human Cytokine kits (Millipore, Billerica, MA). Plate reading will be provided as a fee-for service through Eve Technologies Inc. (Calgary, AB).
Cancer related Symptom Management | At baseline (diagnosis) and then 3, 6, 9, 12 months post diagnosis & every week before and after class during the 12 week intervention
  Participants will complete the ESAS bi-weekly, before and after class. The ESAS is a valid and reliable assessment tool to evaluate the nine more common symptoms experienced by cancer patients (Chang et al., 2000).
Diet Behaviour - 3 Day food record | At baseline (diagnosis) and 4 & 8 weeks, 3, 6, 9, 12 months post diagnosis.
  The 3-Day Diet Record is said to be the most accurate for mean macronutrient content and appropriate for use in studies where subjects may consume a wide variety of foods (American Dietetics Association / Dietitians Canada, 2000). Participants are instructed to record their daily consumption over a period of three days, one of which must be a weekend day. Written instructions and a sample entry are provided to increase accuracy of the daily record.
Diet Behaviour: PG-SGA | At baseline (diagnosis), each week during radiation treatment (6.5 weeks in duration), and 3, 6, 9, 12 months post diagnosis
  The PG-SGA assessment tool has been show to improve treatment outcomes, decrease side-effects, and improve weight-management in cancer patients, and therefore will be used weekly to assess and identify malnutrition among patients (McMahon et al., 2000; Doyle et al., 2006).
Health related Fitness Measures - Resting Heart Rate | At baseline (diagnosis), and 3, 6, 9, 12 months post diagnosis.
  Resting heart rate will be measured by palpating the radial artery and taking a 15 second count as per the CPAFLA protocol (CPAFLA, 2003).
Health Related Fitness Outcome - Blood Pressure | At baseline (diagnosis), and 3, 6, 9, 12 months post diagnosis.
  A resting blood pressure (mmHg) will be measured in duplicate on the left arm using a sphygmomanometer and stethoscope using standardized procedures (CPAFLA, 2003).
Health Related Fitness Outcome - 6 minute walk test | At baseline (diagnosis), and 3, 6, 9, 12 months post diagnosis.
  The six-minute walk test (6MWT) will be used to assess changes in functional aerobic capacity. Using the standardized protocol, participants will be asked to walk as far as they can around a 400-meter track for six minutes [43]. The point reached at 6 minutes will be marked and measured to the nearest 0.5 meter. Rating of perceived exertion (Borg scale) will be completed immediately after completion of the functional aerobic capacity test.
Health Related Fitness Outcome - Grip Strength | At baseline (diagnosis) and 3, 6, 9, and 12 months post diagnosis.
  Muscular strength will be assessed using a combined grip strength of the right and left hands will also be assessed using a hand dynamometer. A sum will be determined in kilograms from the best score of 2 trials recorded for each hand according to the CPAFLA protocol.
Health Related Fitness Outcome - Lower Body Strength | At baseline (diagnosis), and 3, 6, 9, and 12 months post diagnosis
  Lower body strength will be assessed using a 30-second sit to stand test. The number of times participants can stand from a seated position in 30-second will be examined.
Health Related Fitness Outcome - Flexibility | At baseline (diagnosis) and 3, 6, 9, and 12 months post diagnosis
  Flexibility will be assessed by a trunk forward flexion sit-and-reach test using a Wells-Dillon flexometer. The test will follow a standard protocol, with two trials allowed and the highest score to the nearest 0.5 cm recorded.
Health Related Fitness Outcome - Balance | At baseline (diagnosis), and 3, 6, 9, and 12 months post diagnosis.
  Balance will be assessed using a static balance test. The test requires the participant to balance on one foot and then the other as long as they can (length of time to a maximum of 45 seconds) while standing on a 2.54 by 2.54 by 30.5 cm base using a standardized protocol, reported by Fleishman.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Culos-Reed, PhD, Principal Investigator — University of Calgary; Lauren C Capozzi, PhD Student, Study Director — University of Calgary; Harold Lau, MD, Principal Investigator — Tom Baker Cancer Centre, University of Calgary; Raylene Reimer, PhD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Tom Baker Cancer Centre, Calgary, Alberta

REFERENCES:
- [Derived] Capozzi LC, Lau H, Reimer RA, McNeely M, Giese-Davis J, Culos-Reed SN. Exercise and nutrition for head and neck cancer patients: a patient oriented, clinic-supported randomized controlled trial. BMC Cancer. 2012 Oct 2;12:446. doi: 10.1186/1471-2407-12-446. PMID 23031071